CLINICAL TRIAL: NCT00403351
Title: Correlation of Multiple Risk Factors With Presence and Severity of Coronary Artery Disease.
Brief Title: Alternative Risk Markers in Coronary Artery Disease (ARMCAD)
Status: Completed | Type: Observational
Sponsor: Monash University (Other)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other); IM Medical Ltd, Melbourne (Unknown)
Responsible Party: Principal Investigator, Ingrid Hopper, Senior Lecturer, Monash University
Other Study IDs: CP-02/04
Record Dates: First submitted 2006-11-22; First posted 2006-11-23 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Coronary Artery Disease
Keywords: Risk; Coronary artery disease; Heart Rate variability; Pulse wave analysis; BNP; CRP
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum specifically for future cardiac biomarkers
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ARM-CAD 1: Cross-sectional analysis using coronary angiogram results
- ARM-CAD 2: Prospective cohort for incident cardiovascular events and mortality

SUMMARY:
Estimating the risk of future cardiovascular events such as death, stroke and myocardial infarction using traditional risk factors (such as age, gender, smoking, diabetes, hyperlipidaemia and hypertension) is well accepted in patients with and without existing cardiovascular disease. These estimates are based on a number of robust observational studies, including the original Framingham study. While these methods apply reasonably well on a population level their application to the individual patients is not always straightforward. In addition, risk charts, such as those published by the Joint British Societies and American Heart Association, may underestimate risk in certain groups, notably diabetics and patients of Indo-Asian background, whilst overestimating risk in others (by as much as 50% in some studies).

DETAILED DESCRIPTION:
A number of variables including clinical, biochemical, and enzymatic have been evaluated to see if they add to conventional "risk-reduction" models such as Framingham and if so, to understand if they may be used in routine clinical practice.

The aim of this study is to assess several known and a few novel risk-factors (heart rate variability, pulse wave analysis, high-sensitivity CRP and BNP) prior to planned elective coronary angiography (cross-sectional analysis) and in a prospective cohort of high and low-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years or older)
* Male or Female

Exclusion Criteria:

* Acute coronary syndrome
* Urgent angiography
* Assessment would constitute harm to patient
* Informed consent not obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ARM-CAD 1: Patients attending elective coronary angiography ARM-CAD 2: Participants in ARM-CAD 1 plus volunteers with cardiac risk factors
Sampling Method: Non-Probability Sample
Enrollment: 665 (Actual)
Dates: Start 2006-10; Primary Completion 2008-06 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Extent and severity of angiographic coronary artery disease | cross-sectional
All-cause death or myocardial infarction | 1, 2, 5 years
All-cause death, MI or need for cardiac surgery | 1, 2, 5 years

SECONDARY OUTCOMES:
All-cause death | 1, 2, 5 years

OTHER OUTCOMES:
Other cardiovascular events or procedures | 1, 2, 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dipak Kotecha, MB ChB PhD, Principal Investigator — Monash University, Royal Brompton Hospital & University of Birmingham; David Eccleston, MBBS FRACP, Principal Investigator — Monash University and Northern Hospital; Henry Krum, Professor, Principal Investigator — Alfred Hospital / Monash University
Locations (4):
- Australia (4):
  - Box Hill Hospital (Eastern Health), Box Hill, Victoria
  - Caulfield General Medical Centre, Caulfield, Victoria
  - Northern Hospital (Northern Health), Epping, Victoria
  - Alfred Hospital, Melbourne, Victoria

REFERENCES:
- [Result] Kotecha D, Flather M, McGrady M, Pepper J, New G, Krum H, Eccleston D. Contemporary predictors of coronary artery disease in patients referred for angiography. Eur J Cardiovasc Prev Rehabil. 2010 Jun;17(3):280-8. doi: 10.1097/HJR.0b013e3283310108. PMID 19858725
- [Result] Kotecha D, New G, Flather MD, Eccleston D, Pepper J, Krum H. Five-minute heart rate variability can predict obstructive angiographic coronary disease. Heart. 2012 Mar;98(5):395-401. doi: 10.1136/heartjnl-2011-300033. Epub 2011 Nov 25. PMID 22121069
- [Result] Kotecha D, New G, Collins P, Eccleston D, Krum H, Pepper J, Flather MD. Radial artery pulse wave analysis for non-invasive assessment of coronary artery disease. Int J Cardiol. 2013 Aug 10;167(3):917-24. doi: 10.1016/j.ijcard.2012.03.098. Epub 2012 Apr 4. PMID 22483418
- [Derived] Kotecha D, Flather MD, Atar D, Collins P, Pepper J, Jenkins E, Reid CM, Eccleston D; Alternative Risk Markers in Coronary Artery Disease (ARM-CAD) Study. B-type natriuretic peptide trumps other prognostic markers in patients assessed for coronary disease. BMC Med. 2019 Apr 3;17(1):72. doi: 10.1186/s12916-019-1306-9. PMID 30943979
- See also: Study website — http://www.armcad.com